CLINICAL TRIAL: NCT01903681
Title: Open Label, Single Ascending Dose, Cross-over Study to Assess the Pharmacokinetics of Circadin® (Prolonged-Release Melatonin) Mini Tablets in Children With Neurodevelopmental Disorders and Sleep Disturbances
Brief Title: Assessment of the Pharmacokinetics of Circadin® in Children With Neurodevelopmental Disorders and Sleep Disturbances
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Neurim Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: CHDR1219
Record Dates: First submitted 2013-07-16; First posted 2013-07-19 (Estimated); Last update posted 2014-04-04 (Estimated); Status verified 2013-06

CONDITIONS: Sleep Problems
Keywords: Sleep problems, autism spectrum disorder, prolonged-release melatonin, Circadin, endogenous saliva melatonin; Smith-Magenis syndrome, Angelman syndrome, Tuberous Sclerosis
MeSH Terms: conditions — Parasomnias; Autism Spectrum Disorder; Smith-Magenis Syndrome; Angelman Syndrome; Tuberous Sclerosis | interventions — Melatonin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Circadin 10 mg (Active Comparator): Second arm higher dose
  Interventions: Drug: Circadin 10 mg
- Circadin 2 mg (Active Comparator): First arm lower dose
  Interventions: Drug: Circadin 2 mg

INTERVENTIONS:
Drug: Circadin 2 mg — First arm lower dose
  Other Names: non
  Arms: Circadin 2 mg
Drug: Circadin 10 mg — Second arm higher dose
  Arms: Circadin 10 mg

SUMMARY:
There is increasing evidence that chronic sleep disorders in children with autism spectrum disorder (ASD), Angelman Syndrome (AS) and Smith-Magenis syndrome (SMS) are associated with disturbed melatonin secretion and melatonin administration has been shown to be effective in these populations. For children who have difficulties swallowing a tablet, Neurim has developed an age-appropriate Melatonin formulation in the form of mini-tablets which have the same dissolution profile as the Circadin® tablets product, thus should produce the same melatonin concentration-time profile with the same effects. This study concerns the pharmacokinetic study.

The purpose of this study is to :

* Establish the 24 hour baseline profile of endogenous saliva melatonin concentrations and urine 6-SMT excretion in children aged 2 up to and including 17 years with neurodevelopmental disorders with sleep disturbances.
* Establish the concentration-time profile of saliva melatonin concentrations and 24 hour 6-SMT urine excretion after 2 and 10 mg Circadin® mini-tablets single dose administration in children aged 2 up to and including 17 years with neurodevelopmental disorders with sleep disturbances.
* Evaluate the adverse event profile after a single dose of 2 or 10 mg Circadin® mini-tablets in children aged 2 up to and including 17 years with neurodevelopmental disorders with sleep disturbances.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be 2 to 17 years old

Subject has a documented history of autistic spectrum disorder (ASD; as confirmed according to, DSM-IV-TR 299.00, 299.10 and 299.80 or ICD 10: F 84.0, F84.2, F84.3, F84.5, F84.9 ) or one of the following neurogenetic diseases according to ICD 10: Smith-Magenis syndrome, Angelman syndrome or Tuberous Sclerosis (Bourneville's disease)

Subject has current sleep problems; defined as difficulty initiating or maintaining sleep, or non restorative sleep, for at least 1 month (DSM-IV 307.42). Subject is able to comply with taking the study drug and collaborate freely with the study procedures;

Written informed consent from parents having parental responsibility or from the legal guardian(s). In the case of a child is aged 12 years or older the written informed consent of the child is needed in addition to that of parents having responsibility/legal guardian;

Subject is able to understand instructions in Dutch.

Exclusion Criteria:

Subject has history of difficulty with swallowing and/or easy choking;

Subject has current symptoms suggestive of obstructive sleep apnea syndrome or any breathing related sleep disorders or periodic limb movements;

Subject has known clinically significant disturbance(s) in hepatic and/or renal function;

Subject has non-stable epileptic attacks within 3 months prior to screening, in case of a history of epilepsy;

Subject who currently has asthmatic symptoms;

Subject has untreated medical/psychological condition that may be the etiology of sleep disturbances;

Subject is unable to refrain from the use of disallowed concomitant medication ordietary supplements (see paragraph 3.4) from 1 week prior to study occasions;

Subject is unable to refrain from caffeine-containing products for 24 hours before each occasion;

Subject has a known allergy to melatonin;

Female subject who is pregnant at time of screening;

Subject has unstable use of allowed medication within 2 months prior to the screening;

Subject has clinically relevant periodontal disease and/or oral injuries as judged by the investigator;

Subject is unable to refrain from eating bananas and chocolate during the entire day before saliva collection;

Subject is unable to refrain from drinks containing artificial colorants, caffeine (including but not limited to coffee, tea, cola), or alcohol during the day of the collection;

Subject is unable to refrain from aspirin or drugs that contain ibuprofen on the collection day;

Participation in an investigational drug study within 90 days prior to the first dose and/or participation in more than 4 clinical trials in the last year. -

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2013-03; Primary Completion 2014-02 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
baseline profile of endogenous saliva melatonin concentrations and urine 6-SMT excretion | up to 1 year
  To establish the 24 hour baseline profile of endogenous saliva melatonin concentrations and urine 6-SMT excretion in children aged 2 up to and including 17 years with neurodevelopmental disorders with sleep disturbances.
concentration-time profile of saliva melatonin concentrations and 24 hour 6-SMT urine excretion after 2 and 10 mg Circadin® mini-tablets single dose administration | up to 1 year
  To establish the concentration-time profile of saliva melatonin concentrations and 24 hour 6-SMT urine excretion after 2 and 10 mg Circadin® mini-tablets single dose administration in children aged 2 up to and including 17 years with neurodevelopmental disorders with sleep disturbances.
adverse event profile after a single dose of 2 or 10 mg Circadin® mini-tablets | up to 1 year
  To evaluate the adverse event profile after a single dose of 2 or 10 mg Circadin® mini-tablets in children aged 2 up to and including 17 years with neurodevelopmental disorders with sleep disturbances.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Human Drug Research, Leiden, Netherlands